CLINICAL TRIAL: NCT02043379
Title: Intravenous Immunoglobulin for Early Prevention of Cardiopulmonary Bypass Induced Hypogammaglobulinemia in Infants and Neonates
Brief Title: Post-bypass Prophylactic IVIG in Infants and Neonates
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Grifols Biologicals, LLC (Industry)
Responsible Party: Principal Investigator, Jeffrey Alten, MD, Principal Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: F13114002; F13114002 (Other: UAB Institutional Reveiw Board)
Record Dates: First submitted 2014-01-14; First posted 2014-01-23 (Estimated); Results first posted 2017-04-13 (Actual); Last update posted 2017-04-13 (Actual); Status verified 2017-03

CONDITIONS: Hypogammaglobulinemia; Congenital Heart Disease
Keywords: congenital heart disease; Cardiopulmonary Bypass; Hypogammaglobulinemia
MeSH Terms: conditions — Agammaglobulinemia; Heart Defects, Congenital | interventions — Immunoglobulins, Intravenous; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- IVIG (Experimental): Those randomized to the study arm will receive a dose of IVIG 1 gram/kg at 12 hours post-cardiopulmonary bypass. This is a one time only dose and will be administered per hospital standards for IVIG administration.
  Interventions: Drug: IVIG
- Normal Saline (Placebo Comparator): Subject's randomized into the placebo arm of the study will receive a volume of normal saline that is comparative to that if they were to receive IVIG. This will be at 12 hours post-cardiopulmonary bypass. This volume is to ensure blinding of study drug. This infusion will be administered as if the subject is receiving IVIG according to hospital policy.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: IVIG — Those randomized to the study arm will receive a one time dose of IVIG at 12 our post-Cardiopulmonary bypass. This is significantly early than our current standard of care.
  Other Names: Gamunex
  Arms: IVIG
Other: Placebo — If the subject is randomized to the placebo group they will receive a volume of normal saline that is equivalent to the volume of IVIG to be administered based on their weight.
  Other Names: Normal Saline
  Arms: Normal Saline

SUMMARY:
The purpose of this study protocol is to determine if administering Intravenous Immunoglobulin (IVIG) for treatment of cardiopulmonary bypass (CPB) induced hypogammaglobulinemia in the early post-operative period can impact post-surgical outcomes (i.e., infection, fluid overload, and associated morbidities).

DETAILED DESCRIPTION:
The intense post-CPB systemic inflammatory response syndrome (SIRS) is well described in neonates and infants. Increased production and release of pro-inflammatory cytokines, including Tumor Necrosis Factor, Interleukin1-B, and Interleukin-6 may suppress myocardial contractility, induce capillary leak, and activate complement and the clotting cascade - together leading to potential organ injury and death. SIRS is also frequently accompanied by impairment of the humoral immune response. One potential reason for this acquired immunodeficiency after cardiac surgery is the removal of immunoglobulins (Ig)s from the vascular space into other compartments where they are either sequestered or lost from the body altogether. We recently demonstrated that such Ig depletion from the intravascular compartment occurs in neonates following cardiac surgery. In a retrospective study of 53 children <3 months of age, we showed that plasma Immunoglobulin G (IgG) concentration drops precipitously after cardiac surgery and does not return to preoperative levels by 7 days; 51% of patients had hypogammaglobulinemia.

An important question is whether post-CPB low IgG has clinical consequence. IgG plays an essential role in the humoral immune system, activating complement and inducing the phagocytic system to neutralize pathogens. IgG deficiency is a known risk factor for infections in other pediatric populations. We were the first to demonstrate that post-CPB hypogammaglobulinemia is associated with worse clinical outcomes, including increased secondary infections (37% vs.12% in those without low IgG, p<0.05). These novel findings are paramount in that they identify a potential modifiable risk factor to improve outcomes after pediatric cardiac surgery with CPB. Additionally, low IgG is accompanied by fluid overload and prolonged mechanical ventilation. Igs constitute an important component of plasma oncotic pressure, so hypogammaglobulinemia may exacerbate anasarca, prolonging postoperative convalescence and increasing the morbidities associated with increased ICU length of stay.9

Igs have an increasingly recognized role in modulating the innate immune response. Present use of IVIG exceeds mere antibody replacement and extends to the treatment of autoimmune and inflammatory conditions. In fact, more than 75% of IVIG use in the U.S. today is for the treatment of inflammatory conditions, where proposed mechanisms include reduction of pro-inflammatory cytokine and adhesion molecule expression, superantigen neutralization, restoration of glucocorticoid responsiveness, and blockade of complement fragment deposition. It is plausible that IVIG could benefit neonates after cardiac surgery not only via restoration of humoral opsonization capacity, but also as a modulator of innate immunity and SIRS. According to this model, tissue injury, CPB, and shock trigger SIRS, leading to hypogammaglobulinemia and resultant increased susceptibility to inflammatory dysregulation which might be ameliorated via administration of IVIG.

In an adult study, IVIG failed to benefit postoperative cardiac patients with severe SIRS. However, the dose of IVIG given was relatively small compared with that typically given for autoimmune and inflammatory conditions. Neonates and infants may be more susceptible to the harmful effects of acquired hypogammaglobulinemia than adults as they may be unable to generate adequate quantities of antibodies in response to pathogens, relying mainly on maternal Igs until around the 4th to 6th month of life. In addition, they display an exaggerated inflammatory response to CPB as compared with older children and adults, so they might stand to benefit more from IVIG as an immunomodulator.

Because of the increased vulnerability to acquired infection and other morbidities in the setting of hypogammaglobulinemia as result of enhanced SIRS and immune dysfunction, it is feasible that normalization of IgG concentration in the neonatal and infant population may improve clinical outcomes via restoration of the humoral immune system, modulation of the innate immune system, and restoration of intravascular oncotic pressure. The appropriate IgG level threshold for treatment and optimal plasma IgG level to target after administration of IVIG are presently unknown.

ELIGIBILITY:
Inclusion Criteria:

* Infants <6 months old
* Successfully weaned off cardiopulmonary bypass after cardiac surgery

Exclusion Criteria:

* Requirement of extra corporeal membrane oxygenation in the operating room
* Known immune deficiency
* Current Do Not Resuscitate or limitation of care order
* Current enrollment in another interventional clinical study
* Refusal of parental consent

Max Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2014-05; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Alten, MD, Principal Investigator — University of Alabama at Birmingham Pediatric Cardiac Critical Care
Locations (1):
- Children's of Alabama, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared with other individuals

RESULTS

PARTICIPANT FLOW:
Groups:
- IVIG: Those randomized to the study arm will receive a dose of IVIG 1 gram/kg at 12 hours post-cardiopulmonary bypass. This is a one time only dose.
  IVIG: Those randomized to the study arm will receive a one time dose of IVIG at 12 our post-Cardiopulmonary bypass. This is significantly early than our current standard of care.
- Normal Saline: Subject's randomized into the placebo arm of the study will receive a volume of normal saline that is comparative to that if they were to receive IVIG. This will be at 12 hours post-cardiopulmonary bypass. This volume is to ensure blinding of study drug.
  Placebo: If the subject is randomized to the placebo group they will receive a volume of normal saline that is equivalent to the volume of IVIG to be administered based on their weight.
Period: Overall Study
Arm/Group | IVIG | Normal Saline
Started | 30 | 20
Completed | 30 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | IVIG | Normal Saline | Total
Number analyzed (Participants) | 30 | 20 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 30 | 20 | 50
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Inter-Quartile Range); unit: days] | 9 [6 to 50.75] | 47 [6.25 to 79.5] | 11.5 [6 to 74.75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 8 | 22
  Male | 16 | 12 | 28
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 8 | 2 | 10
  White | 22 | 18 | 40
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Weight [Median (Inter-Quartile Range); unit: kilograms] | 3.45 [3.17 to 3.99] | 3.85 [3.04 to 4.52] | 3.51 [3.13 to 4.09]
Gestational Age [Median (Inter-Quartile Range); unit: weeks] | 38 [37 to 39] | 38.5 [37 to 39.75] | 38 [37 to 39]
STAT category [Number; unit: participants] — The Society of Thoracic Surgeons-European Association for Cardio-Thoracic Surgery) Congenital Heart Surgery Mortality Categories. The STAT Mortality Categories range from 1 to 5 with higher values indicating greater risk of mortality associated with operations for congenital heart disease
  participants
    1 | 3 | 0 | 3
    2 | 2 | 5 | 7
    3 | 7 | 8 | 15
    4 | 12 | 4 | 16
    5 | 6 | 3 | 9
Cardiopulmonyar bypass time [Median (Inter-Quartile Range); unit: minutes] | 105.5 [73.5 to 120.3] | 91.5 [68 to 122.3] | 97.5 [70.5 to 120]
Aortic cross clamp time [Median (Inter-Quartile Range); unit: minutes] | 52 [42.5 to 70] | 56 [44.5 to 78.5] | 53.5 [44.5 to 70]
Intubated Pre-operatively [Number; unit: subjects] — Subjects requiring mechanical ventilation in the pre-operative period for either respiratory or cardiac support.
  subjects
    Yes | 5 | 5 | 10
    No | 25 | 15 | 40

OUTCOME MEASURES:

1. Primary Outcome: Post-Operative Infections
Description: The primary endpoint of this study is incidence of post-operative infections through hospital discharge
Time Frame: until Hospital Discharge, an average of 30 days
Measure: Number; unit: subjects
Arm/Group | IVIG | Normal Saline
Number analyzed (Participants) | 30 | 20
subjects
  Yes | 9 | 6
  No | 21 | 14
Statistical Analysis 1: Comparison: IVIG vs Normal Saline; Test type: Non-Inferiority or Equivalence — We used alpha level of 0.05 and power of 0.8 to calculate the sample size necessary to detect a meaningful clinical difference for our primary endpoint; p = 1, Chi-squared — A p-value of <0.05 represents the threshold for statistical significance

2. Primary Outcome: Post-operative Infection
Description: Any positive culture or treatment for culture negative sepsis within 1 week of surgery
Time Frame: within 1 week of surgery
Measure: Number; unit: Subjects
Arm/Group | IVIG | Normal Saline
Number analyzed (Participants) | 30 | 20
Subjects
  Yes | 5 | 3
  No | 25 | 17
Statistical Analysis 1: Comparison: IVIG vs Normal Saline; Test type: Non-Inferiority or Equivalence — Power calculations were not performed on this statistical calculation; p = 1, Chi-squared — A p-value of <0.05 represents the threshold for statistical significance

3. Primary Outcome: Blood Stream Infection
Description: Any positive blood culture during the post-operative period until hospital discharge
Time Frame: until Hospital Discharge, an average of 30 days
Measure: Number; unit: subjects
Arm/Group | IVIG | Normal Saline
Number analyzed (Participants) | 30 | 20
subjects
  Yes | 5 | 1
  No | 25 | 19
Statistical Analysis 1: Comparison: IVIG vs Normal Saline; Test type: Non-Inferiority or Equivalence — Power calculations were not performed on this statistical calculation; p = 0.38, Chi-squared — A p-value of <0.05 represents the threshold for statistical significance

4. Primary Outcome: Blood Stream Infection Within 1 Week of Surgery
Time Frame: 7 days
Measure: Number; unit: subjects
Arm/Group | IVIG | Normal Saline
Number analyzed (Participants) | 30 | 20
subjects
  Yes | 3 | 0
  No | 27 | 20
Statistical Analysis 1: Comparison: IVIG vs Normal Saline; Test type: Non-Inferiority or Equivalence — Power calculations were not performed on this statistical calculation; p = 0.26, Chi-squared — A p-value of <0.05 represents the threshold for statistical significance

5. Secondary Outcome: Post-operative Plasma Albumin
Description: Plasma albumin will be assessed at 24 and 48 hours.
Time Frame: up to 48 hours post CPB
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | IVIG | Normal Saline
Number analyzed (Participants) | 30 | 20
g/dL
  24 hour post-op | 3.7 (0.74) | 4.1 (0.67)
  48 hour post-op | 3.3 (0.57) | 3.6 (0.52)
Statistical Analysis 1: Comparison: IVIG vs Normal Saline; 24 hour post-CPB albumin; Test type: Non-Inferiority or Equivalence — Power calculations were not performed on this statistical calculation; p = 0.42, t-test, 2 sided — A p-value of <0.05 represents the threshold for statistical significance
Statistical Analysis 2: Comparison: IVIG vs Normal Saline; 48 hour post CPB albumin; Test type: Non-Inferiority or Equivalence — Power calculations were not performed on this statistical calculation; p = 0.06, t-test, 2 sided — a p-value of <0.05 represents the threshold for test signficance

6. Secondary Outcome: Fluid Overload Variables
Description: The following fluid overload variables will be assessed in milliliters per kilogram at 0-24 hours post-cardiopulmonary bypass: blood product and albumin administration, chest tube output, urine output, peritoneal dialysis output, net fluid balance, and percent fluid overload. The total output the subject's produce (urine, chest tube, peritoneal drainage, etc.) will be subtracted from the total input (medications, blood products, albumin administration, etc) to determine the total fluid intake in milliliters. This total number will then be divided by the subject's weight in kilograms to determine the fluid overload in mL/kg.
Time Frame: 0-24 hours post-CPB
Measure: Median (Inter-Quartile Range); unit: mililiters/kilogram
Arm/Group | IVIG | Normal Saline
Number analyzed (Participants) | 30 | 20
mililiters/kilogram | 30 [0.6 to 74] | 58.1 [34.4 to 87]
Statistical Analysis 1: Comparison: IVIG vs Normal Saline; Test type: Non-Inferiority or Equivalence — Power calculations were not performed on this statistical calculation; p = 0.52, Wilcoxon (Mann-Whitney) — A p-value of <0.05 represents the threshold for statistical significance

7. Secondary Outcome: Post-operative Inotrope Score
Description: The average admit, 12 hour, 24 hour, and 48 hour post-operative inotrope score will be calculated excluding Milrinone. To calculate the inotrope score the following formula was used: (Epinephrine/Norepinephrine dose in mcg/kg/min x 100) + (Dopamine dose in mcg/kg/min x 1) + (Phenylephrine dose in mcg/kg/min x 10) + (Vasopressin dose unit/kg/hr x 60/10000). The higher the inotrope score the more cardiac support the subject requires. There is not a "normal" scale or range used for this calculation.
Time Frame: first 48 hours post-CPB
Measure: Median (Inter-Quartile Range); unit: inotropic score
Arm/Group | IVIG | Normal Saline
Number analyzed (Participants) | 30 | 20
inotropic score
  Admit | 5 [3.23 to 7.95] | 4.5 [3.15 to 6.6]
  12 hr post-op | 5.3 [3.25 to 7.68] | 5.3 [3 to 8]
  24 hr post-op | 5.3 [3.3 to 7.3] | 5.8 [3.18 to 6.93]
  48 hr post-op | 6.8 [3.08 to 7.83] | 2 [1 to 6.25]
Statistical Analysis 1: Comparison: IVIG vs Normal Saline; Admit Inotrope Score; Test type: Non-Inferiority or Equivalence — Power calculations were not performed on this statistical calculation; p = 0.81, Wilcoxon (Mann-Whitney) — A p-value of <0.05 represents the threshold for statistical significance
Statistical Analysis 2: Comparison: IVIG vs Normal Saline; 12 hours post-operative inotrope score; Test type: Non-Inferiority or Equivalence — power calculations were not performed on this statistical calculation; p = 0.82, Wilcoxon (Mann-Whitney) — a p value of <0.05 represents the threshold for statistical significance
Statistical Analysis 3: Comparison: IVIG vs Normal Saline; 24 hours post-operative inotrope score; Test type: Non-Inferiority or Equivalence — power calculations were not performed on this statistical calculation; p = 0.9, Wilcoxon (Mann-Whitney) — a p value of <0.05 represents the threshold for statistical significance
Statistical Analysis 4: Comparison: IVIG vs Normal Saline; 48 hours post-operative inotrope score; Test type: Non-Inferiority or Equivalence — power calculations were not performed on this statistical calculation; p = 0.23, Wilcoxon (Mann-Whitney) — a p-value of <0.05 represents the threshold for statistical signficance

8. Secondary Outcome: Respiratory Variables
Description: Alive, ventilator free days will be recorded at hospital discharge.
Time Frame: until Hospital Discharge, an average of 30 days
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | IVIG | Normal Saline
Number analyzed (Participants) | 30 | 20
days | 24.7 [21.1 to 26.3] | 25.5 [21.6 to 27]
Statistical Analysis 1: Comparison: IVIG vs Normal Saline; Test type: Non-Inferiority or Equivalence — Power calculations were not performed on this statistical calculation; p = 0.49, Wilcoxon (Mann-Whitney) — A p-value of <0.05 represents the threshold for statistical significance

9. Secondary Outcome: Hospital Discharge
Description: From admit post-operative to the Pediatric cardiac intensive care unit until discharge from the hospital in days.
Time Frame: Approximately 1 month
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | IVIG | Normal Saline
Number analyzed (Participants) | 30 | 20
days | 22 [11.25 to 35] | 22 [7.25 to 34.75]
Statistical Analysis 1: Comparison: IVIG vs Normal Saline; Test type: Non-Inferiority or Equivalence — Power calculations were not performed on this statistical calculation; p = 0.79, Wilcoxon (Mann-Whitney) — A p-value of <0.05 represents the threshold for statistical significance

10. Secondary Outcome: Plasma Immunoglobulins
Description: Plasma Immunoglobulin levels will be checked pre-operatively, 12 hours post-op and 5 days post-op
Time Frame: 5 days post-op
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | IVIG | Normal Saline
Number analyzed (Participants) | 30 | 20
mg/dL
  Pre-operative serum IgG level | 487 (226.1) | 414 (230.5)
  12 hour post-operative serum IgG level | 496 (183) | 569 (272)
  Post-operative day 3 serum IgG level | 837 (243) | 508 (215.4)
  Post-operative day 5 serum IgG level | 839 (213) | 585 (212.3)
Statistical Analysis 1: Comparison: IVIG vs Normal Saline; pre-operative IgG level; Test type: Non-Inferiority or Equivalence — Power calculations were not performed on this statistical calculation; p = 0.32, t-test, 2 sided — A p-value of <0.05 represents the threshold for statistical significance
Statistical Analysis 2: Comparison: IVIG vs Normal Saline; 12 hours post-operative IgG level; Test type: Non-Inferiority or Equivalence — power calculations were not performed on this statistical calculation; p = 0.36, Wilcoxon (Mann-Whitney) — a p-value of <0.05 represents the threshold for statistical significance
Statistical Analysis 3: Comparison: IVIG vs Normal Saline; post-operative day 3 (72 hours) IgG level; Test type: Non-Inferiority or Equivalence — power calculations were not performed on this statistical calculation; p < 0.01, Wilcoxon (Mann-Whitney) — p-value of <0.05 represents the threshold for statistical signficance
Statistical Analysis 4: Comparison: IVIG vs Normal Saline; post-operative day 5 (120 hours) IgG level; Test type: Non-Inferiority or Equivalence — power calculations were not performed on this statistical calculation; p < 0.01, Wilcoxon (Mann-Whitney) — p-value of <0.05 represents the threshold for statistical significance

11. Secondary Outcome: Interferon-gamma Plasma Cytokine Levels
Description: Plasma cytokine levels measured preoperatively, 0, 4, 12, 24 hours, and 48 hours post-operatively.
Time Frame: Pre-operative to 48 hours post-operative
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | IVIG | Normal Saline
Number analyzed (Participants) | 30 | 20
pg/mL
  Pre-operative | 2.2 [0.7 to 4.5] | 3.5 [2.5 to 7.7]
  0 hour post-op | 2.6 [1.3 to 4.2] | 6 [3.4 to 12.4]
  4 hour post-op | 2.8 [2.2 to 4.1] | 6.1 [3 to 16]
  12 hour post-op | 2.8 [2 to 4.5] | 6.3 [2.6 to 10.4]
  24 hour post-op | 2 [1.3 to 3.2] | 5.6 [2.7 to 11.5]
  48 hour post-op | 2.2 [1.4 to 3.2] | 3.4 [2.3 to 5.2]
Statistical Analysis 1: Comparison: IVIG vs Normal Saline; pre-operative; Test type: Non-Inferiority or Equivalence — Power calculations were not performed on this statistical calculation; p = 0.60, Wilcoxon (Mann-Whitney) — A p-value of <0.05 represents the threshold for statistical significance
Statistical Analysis 2: Comparison: IVIG vs Normal Saline; 0 hour post-operative; Test type: Non-Inferiority or Equivalence — Power calculations were not performed on this statistical calculation; p = 0.06, Wilcoxon (Mann-Whitney) — A p-value of <0.05 represents the threshold for statistical significance
Statistical Analysis 3: Comparison: IVIG vs Normal Saline; 4 hour post-operative; Test type: Non-Inferiority or Equivalence — Power calculations were not performed on this statistical calculation; p = 0.06, Wilcoxon (Mann-Whitney) — A p-value of <0.05 represents the threshold for statistical significance
Statistical Analysis 4: Comparison: IVIG vs Normal Saline; 12 hours post-operative; Test type: Non-Inferiority or Equivalence — Power calculations were not performed on this statistical calculation; p = 0.33, Wilcoxon (Mann-Whitney) — A p-value of <0.05 represents the threshold for statistical significance
Statistical Analysis 5: Comparison: IVIG vs Normal Saline; 24 hours post-operative; Test type: Non-Inferiority or Equivalence — Power calculations were not performed on this statistical calculation; p = 0.05, Wilcoxon (Mann-Whitney) — A p-value of <0.05 represents the threshold for statistical significance
Statistical Analysis 6: Comparison: IVIG vs Normal Saline; 48 hours post-operative; Test type: Non-Inferiority or Equivalence — Power calculations were not performed on this statistical calculation; p = 0.83, Wilcoxon (Mann-Whitney) — A p-value of <0.05 represents the threshold for statistical significance

12. Secondary Outcome: Immunoglobulin Concentration in Chest Tube Drainage
Description: Immunoglobulin concentration will be measured from chest tube every 4 hours for first 12 hours post-operative and then 24 hours post-operative.
Time Frame: 24 hours post-op
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | IVIG | Normal Saline
Number analyzed (Participants) | 30 | 20
mg/dL
  0 hr post-op | 50.9 [23.3 to 73.6] | 62.2 [39.4 to 117.5]
  4 hr post-op | 154.3 [79.4 to 250.7] | 161.3 [111 to 291.2]
  8 hr post-op | 195.2 [122.3 to 308.6] | 227.6 [150.6 to 448.1]
  12 hr post-op | 233.5 [155.3 to 316.3] | 226.8 [202.4 to 447.2]
  24 hr post-op | 614.2 [471 to 916.4] | 268.7 [190.1 to 578]
Statistical Analysis 1: Comparison: IVIG vs Normal Saline; 0 hour levels; Test type: Non-Inferiority or Equivalence — Power calculations were not performed on this statistical calculation; p = 0.27, Wilcoxon (Mann-Whitney) — A p-value of <0.05 represents the threshold for statistical significance
Statistical Analysis 2: Comparison: IVIG vs Normal Saline; 4 hour level; Test type: Non-Inferiority or Equivalence — Power calculations were not performed on this statistical calculation; p = 0.34, Wilcoxon (Mann-Whitney) — A p-value of <0.05 represents the threshold for statistical significance
Statistical Analysis 3: Comparison: IVIG vs Normal Saline; 8 hour level; Test type: Non-Inferiority or Equivalence — Power calculations were not performed on this statistical calculation; p = 0.14, Wilcoxon (Mann-Whitney) — A p-value of <0.05 represents the threshold for statistical significance
Statistical Analysis 4: Comparison: IVIG vs Normal Saline; 12 hour level; Test type: Non-Inferiority or Equivalence — Power calculations were not performed on this statistical calculation; p = 0.13, Wilcoxon (Mann-Whitney) — A p-value of <0.05 represents the threshold for statistical significance
Statistical Analysis 5: Comparison: IVIG vs Normal Saline; 24 hour level; Test type: Non-Inferiority or Equivalence — Power calculations were not performed on this statistical calculation; p = 0.02, Wilcoxon (Mann-Whitney) — A p-value of <0.05 represents the threshold for statistical significance

13. Secondary Outcome: Mortality
Description: Incidence of mortality from admit to Pediatric cardiac intensive care unit post-operatively until hospital discharge .
Time Frame: Approximately 1 month
Measure: Number; unit: subjects
Arm/Group | IVIG | Normal Saline
Number analyzed (Participants) | 30 | 20
subjects
  Yes | 3 | 2
  No | 27 | 18
Statistical Analysis 1: Comparison: IVIG vs Normal Saline; Test type: Non-Inferiority or Equivalence — Power calculations were not performed on this statistical calculation; p = 1, Chi-squared — A p-value of <0.05 represents the threshold for statistical significance

14. Secondary Outcome: Intensive Care Unit Length of Stay
Description: The length of stay in the pediatric cardiac intensive care unit from admit post-operative until either discharge home, discharge to another unit/hospital/care facility, or death. This value is calculated in hours. Admit post-operative is recorded as hour 0.
Time Frame: 1 month
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | IVIG | Normal Saline
Number analyzed (Participants) | 30 | 20
hours | 357.9 [141.3 to 536.6] | 189.6 [106.0 to 575.8]
Statistical Analysis 1: Comparison: IVIG vs Normal Saline; Test type: Non-Inferiority or Equivalence — Power calculations were not performed on this statistical calculation; p = 0.4, Wilcoxon (Mann-Whitney) — A p-value of <0.05 represents the threshold for statistical significance

15. Secondary Outcome: Fluid Overload Variables
Description: The following fluid overload variables will be assessed at 0-24 hours, 25-48 hours, and 0-48 hours post-cardiopulmonary bypass: blood product and albumin administration, chest tube output, urine output, peritoneal dialysis output, net fluid balance, and percent fluid overload.The total output the subject's produce (urine, chest tube, peritoneal drainage, etc.) will be subtracted from the total input (medications, blood products, albumin administration, etc) to determine the total fluid intake in milliliters. This total number will then be divided by the subject's weight in kilograms to determine the fluid overload in mL/kg.
Time Frame: 0-48 hours post-CPB
Measure: Median (Inter-Quartile Range); unit: militers/kilogram
Arm/Group | IVIG | Normal Saline
Number analyzed (Participants) | 30 | 20
militers/kilogram
  0-24 hours post-CPB | 30 [0.6 to 74] | 58.1 [34.4 to 87]
  25-48 hours post-CPB | 7.4 [-35.53 to 41.55] | 34.9 [-0.4 to 43.85]
  0-48 hours post-CPB | 46.6 [13.9 to 85.25] | 77 [36.8 to 114.73]
Statistical Analysis 1: Comparison: IVIG vs Normal Saline; 0-48 hours post-CPB; Test type: Non-Inferiority or Equivalence — Power calculations were not performed on this statistical calculation; p = 0.09, Wilcoxon (Mann-Whitney) — A p-value of <0.05 represents the threshold for statistical significance
Statistical Analysis 2: Comparison: IVIG vs Normal Saline; 0-24 hours post CPB; Test type: Non-Inferiority or Equivalence — Power calculations were not performed on this statistical calculation; p = 0.52, Wilcoxon (Mann-Whitney) — A p-value of <0.05 represents the threshold for statistical significance

16. Secondary Outcome: Respiratory Variables
Description: Time until first extubation in hours
Time Frame: until extubation, an average of 2 days
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | IVIG | Normal Saline
Number analyzed (Participants) | 30 | 20
hours | 46 [18.5 to 88.1] | 43 [18 to 93.2]
Statistical Analysis 1: Comparison: IVIG vs Normal Saline; Test type: Non-Inferiority or Equivalence — Power calculations were not performed on this statistical calculation; p = 0.72, Wilcoxon (Mann-Whitney) — A p-value of <0.05 represents the threshold for statistical significance

17. Secondary Outcome: Respiratory Variables
Description: Total time duration of post-operative length of mechanical ventilation until hospital discharge
Time Frame: until extubation, an average of 2 days
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | IVIG | Normal Saline
Number analyzed (Participants) | 30 | 20
hours | 62.1 [29.9 to 165] | 59 [23.3 to 153.5]
Statistical Analysis 1: Comparison: IVIG vs Normal Saline; Test type: Non-Inferiority or Equivalence — Power calculations were not performed on this statistical calculation; p = 0.63, Wilcoxon (Mann-Whitney) — A p-value of <0.05 represents the threshold for statistical significance

18. Secondary Outcome: Interleukin-10 Plasma Cytokine Levels
Description: Plasma cytokine levels measured preoperatively, 0, 4, 12, 24 hours, and 48 hours post-operatively.
Time Frame: pre-operative through 48 hours post-operative
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | IVIG | Normal Saline
Number analyzed (Participants) | 30 | 20
pg/mL
  Pre-operative | 1.4 [1 to 3.2] | 1.8 [1.1 to 3]
  0 hour post-operative | 54.4 [37.5 to 91.7] | 124 [52.5 to 216.5]
  4 hour post-operative | 10.1 [6.4 to 25.3] | 20.1 [7.9 to 56.7]
  12 hour post-operative | 4.7 [2.7 to 7.9] | 10.2 [5.5 to 20.9]
  24 hour post-operative | 1.8 [1.2 to 3.6] | 4 [2 to 6.7]
  48 hour post-operatiave | 1.1 [0.8 to 2.3] | 2.3 [1.2 to 9.8]
Statistical Analysis 1: Comparison: IVIG vs Normal Saline; pre-operative; Test type: Non-Inferiority or Equivalence — Power calculations were not performed on this statistical calculation; p = 0.41, Wilcoxon (Mann-Whitney) — A p-value of <0.05 represents the threshold for statistical significance
Statistical Analysis 2: Comparison: IVIG vs Normal Saline; 0 hour post-operative; Test type: Non-Inferiority or Equivalence — Power calculations were not performed on this statistical calculation; p = 0.34, Wilcoxon (Mann-Whitney) — A p-value of <0.05 represents the threshold for statistical significance
Statistical Analysis 3: Comparison: IVIG vs Normal Saline; 4 hour post-operative; Test type: Non-Inferiority or Equivalence — Power calculations were not performed on this statistical calculation; p = 0.47, Wilcoxon (Mann-Whitney) — A p-value of <0.05 represents the threshold for statistical significance
Statistical Analysis 4: Comparison: IVIG vs Normal Saline; 12 hour post-operative; Test type: Non-Inferiority or Equivalence — Power calculations were not performed on this statistical calculation; p = 0.42, Wilcoxon (Mann-Whitney) — A p-value of <0.05 represents the threshold for statistical significance
Statistical Analysis 5: Comparison: IVIG vs Normal Saline; 24 hour post-operative; Test type: Non-Inferiority or Equivalence — Power calculations were not performed on this statistical calculation; p = 0.82, Wilcoxon (Mann-Whitney) — A p-value of <0.05 represents the threshold for statistical significance
Statistical Analysis 6: Comparison: IVIG vs Normal Saline; 48 hour post-operative; Test type: Non-Inferiority or Equivalence — Power calculations were not performed on this statistical calculation; p = 0.44, Wilcoxon (Mann-Whitney) — A p-value of <0.05 represents the threshold for statistical significance

19. Secondary Outcome: Interleukin-12p70 Plasma Cytokine Levels
Description: Plasma cytokine levels measured preoperatively, 0, 4, 12, 24 hours, and 48 hours post-operatively.
Time Frame: pre-operative through 48 hours post-operative
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | IVIG | Normal Saline
Number analyzed (Participants) | 30 | 20
pg/mL
  Pre-operative | 0.2 [0.2 to 0.2] | 0.2 [0.2 to 0.6]
  0 hour post-operative | 0.2 [0.2 to 0.3] | 0.6 [0.3 to 2.1]
  4 hour post-operative | 0.4 [0.3 to 0.5] | 0.5 [0.3 to 3.5]
  12 hour post-operative | 0.5 [0.3 to 0.8] | 1 [0.4 to 2]
  24 hour post-operative | 0.3 [0.2 to 0.5] | 0.7 [0.3 to 1.6]
  48 hour post-operatiave | 0.2 [0.2 to 0.3] | 0.4 [0.2 to 0.8]
Statistical Analysis 1: Comparison: IVIG vs Normal Saline; pre-operative; Test type: Non-Inferiority or Equivalence — Power calculations were not performed on this statistical calculation; p = 0.28, Wilcoxon (Mann-Whitney) — A p-value of <0.05 represents the threshold for statistical significance
Statistical Analysis 2: Comparison: IVIG vs Normal Saline; 0 hour post-operative; Test type: Non-Inferiority or Equivalence — Power calculations were not performed on this statistical calculation; p = 0.37, Wilcoxon (Mann-Whitney) — A p-value of <0.05 represents the threshold for statistical significance
Statistical Analysis 3: Comparison: IVIG vs Normal Saline; 4 hour post-operative; Test type: Non-Inferiority or Equivalence — Power calculations were not performed on this statistical calculation; p = 0.42, Wilcoxon (Mann-Whitney) — A p-value of <0.05 represents the threshold for statistical significance
Statistical Analysis 4: Comparison: IVIG vs Normal Saline; 12 hour post-operative; Test type: Non-Inferiority or Equivalence — Power calculations were not performed on this statistical calculation; p = 0.31, Wilcoxon (Mann-Whitney) — A p-value of <0.05 represents the threshold for statistical significance
Statistical Analysis 5: Comparison: IVIG vs Normal Saline; 24 hour post-operative; Test type: Non-Inferiority or Equivalence — Power calculations were not performed on this statistical calculation; p = 0.38, Wilcoxon (Mann-Whitney) — A p-value of <0.05 represents the threshold for statistical significance
Statistical Analysis 6: Comparison: IVIG vs Normal Saline; 48 hour post-operative; Test type: Non-Inferiority or Equivalence — Power calculations were not performed on this statistical calculation; p = 0.4, Wilcoxon (Mann-Whitney) — A p-value of <0.05 represents the threshold for statistical significance

20. Secondary Outcome: Interleukin-1b Plasma Cytokine Levels
Description: Plasma cytokine levels measured preoperatively, 0, 4, 12, 24 hours, and 48 hours post-operatively.
Time Frame: pre-operative through 48 hours post-operative
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | IVIG | Normal Saline
Number analyzed (Participants) | 30 | 20
pg/mL
  Pre-operative | 0.2 [0.1 to 0.2] | 0.2 [0.1 to 0.7]
  0 hour post-operative | 0.3 [0.2 to 0.4] | 0.4 [0.3 to 0.4]
  4 hour post-operative | 0.3 [0.3 to 0.6] | 0.5 [0.4 to 0.6]
  12 hour post-operative | 0.3 [0.3 to 0.5] | 0.3 [0.2 to 0.3]
  24 hour post-operative | 0.3 [0.2 to 0.5] | 0.5 [0.3 to 1.4]
  48 hour post-operatiave | 0.3 [0.2 to 0.6] | 0.3 [0.2 to 0.4]
Statistical Analysis 1: Comparison: IVIG vs Normal Saline; pre-operative; Test type: Non-Inferiority or Equivalence — Power calculations were not performed on this statistical calculation; p = 0.1, Wilcoxon (Mann-Whitney) — A p-value of <0.05 represents the threshold for statistical significance
Statistical Analysis 2: Comparison: IVIG vs Normal Saline; 0 hour post-operative; Test type: Non-Inferiority or Equivalence — Power calculations were not performed on this statistical calculation; p = 0.12, Wilcoxon (Mann-Whitney) — A p-value of <0.05 represents the threshold for statistical significance
Statistical Analysis 3: Comparison: IVIG vs Normal Saline; 4 hour post-operative; Test type: Non-Inferiority or Equivalence — Power calculations were not performed on this statistical calculation; p = 0.51, Wilcoxon (Mann-Whitney) — A p-value of <0.05 represents the threshold for statistical significance
Statistical Analysis 4: Comparison: IVIG vs Normal Saline; 12 hour post-operative; Test type: Non-Inferiority or Equivalence — Power calculations were not performed on this statistical calculation; p = 0.27, Wilcoxon (Mann-Whitney) — A p-value of <0.05 represents the threshold for statistical significance
Statistical Analysis 5: Comparison: IVIG vs Normal Saline; 24 hour post-operative; Test type: Non-Inferiority or Equivalence — Power calculations were not performed on this statistical calculation; p = 0.88, Wilcoxon (Mann-Whitney) — A p-value of <0.05 represents the threshold for statistical significance
Statistical Analysis 6: Comparison: IVIG vs Normal Saline; 48 hour post-operative; Test type: Non-Inferiority or Equivalence — Power calculations were not performed on this statistical calculation; p = 0.38, Wilcoxon (Mann-Whitney) — A p-value of <0.05 represents the threshold for statistical significance

21. Secondary Outcome: Interleukin-6 Plasma Cytokine Levels
Description: Plasma cytokine levels measured preoperatively, 0, 4, 12, 24 hours, and 48 hours post-operatively.
Time Frame: pre-operative through 48 hours post-operative
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | IVIG | Normal Saline
Number analyzed (Participants) | 30 | 20
pg/mL
  Pre-operative | 2.1 [1.1 to 5.5] | 3.3 [1.4 to 7.6]
  0 hour post-operative | 10.3 [6.6 to 16.2] | 17.3 [9.9 to 30.7]
  4 hour post-operative | 32.6 [23.6 to 46.5] | 52.4 [33.8 to 84.9]
  12 hour post-operative | 43.6 [29.6 to 64.8] | 49.8 [36.6 to 86.6]
  24 hour post-operative | 26.3 [15.6 to 50.4] | 40.8 [24.2 to 81.3]
  48 hour post-operatiave | 15.8 [9.4 to 21.5] | 15.5 [10.5 to 24.8]
Statistical Analysis 1: Comparison: IVIG vs Normal Saline; pre-operative; Test type: Non-Inferiority or Equivalence — Power calculations were not performed on this statistical calculation; p = 0.35, Wilcoxon (Mann-Whitney) — A p-value of <0.05 represents the threshold for statistical significance
Statistical Analysis 2: Comparison: IVIG vs Normal Saline; 0 hour post-operative; Test type: Non-Inferiority or Equivalence — Power calculations were not performed on this statistical calculation; p = 0.39, Wilcoxon (Mann-Whitney) — A p-value of <0.05 represents the threshold for statistical significance
Statistical Analysis 3: Comparison: IVIG vs Normal Saline; 4 hour post-operative; Test type: Non-Inferiority or Equivalence — Power calculations were not performed on this statistical calculation; p = 0.58, Wilcoxon (Mann-Whitney) — A p-value of <0.05 represents the threshold for statistical significance
Statistical Analysis 4: Comparison: IVIG vs Normal Saline; 12 hour post-operative; Test type: Non-Inferiority or Equivalence — Power calculations were not performed on this statistical calculation; p = 0.36, Wilcoxon (Mann-Whitney) — A p-value of <0.05 represents the threshold for statistical significance
Statistical Analysis 5: Comparison: IVIG vs Normal Saline; 24 hour post-operative; Test type: Non-Inferiority or Equivalence — Power calculations were not performed on this statistical calculation; p = 0.61, Wilcoxon (Mann-Whitney) — A p-value of <0.05 represents the threshold for statistical significance
Statistical Analysis 6: Comparison: IVIG vs Normal Saline; 48 hour post-operative; Test type: Non-Inferiority or Equivalence — Power calculations were not performed on this statistical calculation; p = 0.38, Wilcoxon (Mann-Whitney) — A p-value of <0.05 represents the threshold for statistical significance

22. Secondary Outcome: Interleukin-8 Plasma Cytokine Levels
Description: Plasma cytokine levels measured preoperatively, 0, 4, 12, 24 hours, and 48 hours post-operatively.
Time Frame: pre-operative through 48 hours post-operative
Measure: Median (Inter-Quartile Range); unit: pg/dL
Arm/Group | IVIG | Normal Saline
Number analyzed (Participants) | 30 | 20
pg/dL
  Pre-operative | 18.7 [14.4 to 22.7] | 17.7 [12.8 to 23.4]
  0 hour post-operative | 76.5 [58.8 to 131] | 163 [99.9 to 255.5]
  4 hour post-operative | 116.5 [63.6 to 162.3] | 147.5 [71 to 214.8]
  12 hour post-operative | 67.1 [36.7 to 131] | 90 [50 to 132]
  24 hour post-operative | 47.7 [40.3 to 61.7] | 46 [33.4 to 112.8]
  48 hour post-operatiave | 33.6 [24.6 to 59.8] | 38.2 [23.6 to 64.7]
Statistical Analysis 1: Comparison: IVIG vs Normal Saline; pre-operative; Test type: Non-Inferiority or Equivalence — Power calculations were not performed on this statistical calculation; p = 0.1, Wilcoxon (Mann-Whitney) — A p-value of <0.05 represents the threshold for statistical significance
Statistical Analysis 2: Comparison: IVIG vs Normal Saline; 0 hour post-operative; Test type: Non-Inferiority or Equivalence — Power calculations were not performed on this statistical calculation; p = 0.02, Wilcoxon (Mann-Whitney) — A p-value of <0.05 represents the threshold for statistical significance
Statistical Analysis 3: Comparison: IVIG vs Normal Saline; 4 hour post-operative; Test type: Non-Inferiority or Equivalence — Power calculations were not performed on this statistical calculation; p = 0.34, Wilcoxon (Mann-Whitney) — A p-value of <0.05 represents the threshold for statistical significance
Statistical Analysis 4: Comparison: IVIG vs Normal Saline; 12 hour post-operative; Test type: Non-Inferiority or Equivalence — Power calculations were not performed on this statistical calculation; p = 0.35, Wilcoxon (Mann-Whitney) — A p-value of <0.05 represents the threshold for statistical significance
Statistical Analysis 5: Comparison: IVIG vs Normal Saline; 24 hour post-operative; Test type: Non-Inferiority or Equivalence — Power calculations were not performed on this statistical calculation; p = 0.67, Wilcoxon (Mann-Whitney) — A p-value of <0.05 represents the threshold for statistical significance
Statistical Analysis 6: Comparison: IVIG vs Normal Saline; 48 hour post-operative; Test type: Non-Inferiority or Equivalence — Power calculations were not performed on this statistical calculation; p = 0.47, Wilcoxon (Mann-Whitney) — A p-value of <0.05 represents the threshold for statistical significance

23. Secondary Outcome: Tumor Necrosis Factor Plasma Cytokine Levels
Description: Plasma cytokine levels measured preoperatively, 0, 4, 12, 24 hours, and 48 hours post-operatively.
Time Frame: pre-operative through 48 hours post-operative
Measure: Median (Inter-Quartile Range); unit: pg/dL
Arm/Group | IVIG | Normal Saline
Number analyzed (Participants) | 30 | 20
pg/dL
  Pre-operative | 2.3 [1.9 to 3.4] | 2.9 [2.4 to 4]
  0 hour post-operative | 2.9 [2.2 to 3.8] | 4.3 [2.5 to 6.4]
  4 hour post-operative | 3.7 [2.6 to 5.6] | 5.3 [3.7 to 7.6]
  12 hour post-operative | 3.1 [2.2 to 3.4] | 4.1 [2.7 to 5.5]
  24 hour post-operative | 2.9 [2.2 to 3.4] | 3.8 [3 to 5]
  48 hour post-operatiave | 2.4 [2 to 3.2] | 3.5 [2.1 to 4.8]
Statistical Analysis 1: Comparison: IVIG vs Normal Saline; pre-operative; Test type: Non-Inferiority or Equivalence — Power calculations were not performed on this statistical calculation; p = 0.46, Wilcoxon (Mann-Whitney) — A p-value of <0.05 represents the threshold for statistical significance
Statistical Analysis 2: Comparison: IVIG vs Normal Saline; 0 hour post-operative; Test type: Non-Inferiority or Equivalence — Power calculations were not performed on this statistical calculation; p = 0.04, Wilcoxon (Mann-Whitney) — A p-value of <0.05 represents the threshold for statistical significance
Statistical Analysis 3: Comparison: IVIG vs Normal Saline; 4 hour post-operative; Test type: Non-Inferiority or Equivalence — Power calculations were not performed on this statistical calculation; p = 0.14, Wilcoxon (Mann-Whitney) — A p-value of <0.05 represents the threshold for statistical significance
Statistical Analysis 4: Comparison: IVIG vs Normal Saline; 12 hour post-operative; Test type: Non-Inferiority or Equivalence — Power calculations were not performed on this statistical calculation; p = 0.82, Wilcoxon (Mann-Whitney) — A p-value of <0.05 represents the threshold for statistical significance
Statistical Analysis 5: Comparison: IVIG vs Normal Saline; 24 hour post-operative; Test type: Non-Inferiority or Equivalence — Power calculations were not performed on this statistical calculation; p = 0.9, Wilcoxon (Mann-Whitney) — A p-value of <0.05 represents the threshold for statistical significance
Statistical Analysis 6: Comparison: IVIG vs Normal Saline; 48 hour post-operative; Test type: Non-Inferiority or Equivalence — Power calculations were not performed on this statistical calculation; p = 0.78, Wilcoxon (Mann-Whitney) — A p-value of <0.05 represents the threshold for statistical significance

24. Secondary Outcome: Immunoglobulin Concentration in Peritoneal Dialysis Drainage
Description: Immunoglobulin concentration will be measured from chest tube and peritoneal drain every 4 hours for first 12 hours post-operative and 24 hours post-operative.
Time Frame: 24 hours post-op
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | IVIG | Normal Saline
Number analyzed (Participants) | 30 | 20
mg/dL
  0 hr post-op | 33.1 [18.8 to 52.1] | 101.6 [11.5 to 144.3]
  4 hr post-op | 136.2 [45.6 to 263.3] | 201.6 [114.5 to 384.2]
  8 hr post-op | 279.8 [193.4 to 446.8] | 221.2 [84.4 to 513.2]
  12 hr post-op | 387.33 [143.1 to 510.2] | 300.1 [149.4 to 434.3]
  24 hr post-op | 1613.9 [598.3 to 2181.1] | 366.9 [170.4 to 984.2]
Statistical Analysis 1: Comparison: IVIG vs Normal Saline; 0 hour level; Test type: Non-Inferiority or Equivalence — Power calculations were not performed on this statistical calculation; p = 0.37, Wilcoxon (Mann-Whitney) — A p-value of <0.05 represents the threshold for statistical significance
Statistical Analysis 2: Comparison: IVIG vs Normal Saline; 4 hour level; Test type: Non-Inferiority or Equivalence — Power calculations were not performed on this statistical calculation; p = 0.47, Wilcoxon (Mann-Whitney) — A p-value of <0.05 represents the threshold for statistical significance
Statistical Analysis 3: Comparison: IVIG vs Normal Saline; 8 hour level; Test type: Non-Inferiority or Equivalence — Power calculations were not performed on this statistical calculation; p = 0.47, Wilcoxon (Mann-Whitney) — A p-value of <0.05 represents the threshold for statistical significance
Statistical Analysis 4: Comparison: IVIG vs Normal Saline; 12 hour level; Test type: Non-Inferiority or Equivalence — Power calculations were not performed on this statistical calculation; p = 0.79, Wilcoxon (Mann-Whitney) — A p-value of <0.05 represents the threshold for statistical significance
Statistical Analysis 5: Comparison: IVIG vs Normal Saline; 24 hour level; Test type: Non-Inferiority or Equivalence — Power calculations were not performed on this statistical calculation; p = 0.04, Wilcoxon (Mann-Whitney) — A p-value of <0.05 represents the threshold for statistical significance

25. Secondary Outcome: Serum Creatinine
Description: Pre-operative and 48 hour post-operative maximum creatinine recorded.
Time Frame: 48 hours
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | IVIG | Normal Saline
Number analyzed (Participants) | 30 | 20
mg/dL
  Pre-operative | 0.4 (0.15) | 0.4 (0.17)
  Max | 0.8 (0.28) | 0.7 (0.38)
Statistical Analysis 1: Comparison: IVIG vs Normal Saline; pre-operative; Test type: Non-Inferiority or Equivalence — Power calculations were not performed on this statistical calculation; p = 0.43, t-test, 2 sided — A p-value of <0.05 represents the threshold for statistical significance
Statistical Analysis 2: Comparison: IVIG vs Normal Saline; max; Test type: Non-Inferiority or Equivalence — Power calculations were not performed on this statistical calculation; p = 0.68, t-test, 2 sided — A p-value of <0.05 represents the threshold for statistical significance

26. Secondary Outcome: Lactic Acid
Time Frame: pre-operative through 24 hours post-operative
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | IVIG | Normal Saline
Number analyzed (Participants) | 30 | 20
mmol/L
  Pre-operative | 1.3 (0.65) | 1.4 (0.75)
  24 hour maximum | 5.7 (4) | 5.4 (4.54)
Statistical Analysis 1: Comparison: IVIG vs Normal Saline; pre-operative; Test type: Non-Inferiority or Equivalence — Power calculations were not performed on this statistical calculation; p = 0.87, t-test, 2 sided — A p-value of <0.05 represents the threshold for statistical significance
Statistical Analysis 2: Comparison: IVIG vs Normal Saline; 24 hour post-operative max; Test type: Non-Inferiority or Equivalence — Power calculations were not performed on this statistical calculation; p = 0.79, t-test, 2 sided — A p-value of <0.05 represents the threshold for statistical significance

ADVERSE EVENTS:
Arm/Group | IVIG | Normal Saline
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/20
Other Adverse Events (participants affected / at risk) | 0/30 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes